CLINICAL TRIAL: NCT01926041
Title: The Effectiveness of Smoking Cessation in Prediabetic Smokers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201303041RINB
Record Dates: First submitted 2013-08-06; First posted 2013-08-20 (Estimated); Results first posted 2023-02-22 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus; Cigarette Smoking; Prediabetes
Keywords: community; preventive medicine; prediabetes; smoking cessation
MeSH Terms: conditions — Diabetes Mellitus; Cigarette Smoking; Prediabetic State; Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): A 16-week FIT2 program that combines smoking cessation therapy with individualized behavior coaching in diet and physical activity for PCWG restriction.
  Interventions: Drug: Varenicline for tobacco smoking cessation; Behavioral: Individualized counseling about both smoking cessation and weight control techniques
- Control (No Intervention): Usual care

INTERVENTIONS:
Drug: Varenicline for tobacco smoking cessation — The 16-week varenicline course conforms to real-practice government regulations in Taiwan.
  Other Names: Varenicline (Champix)
  Arms: Intervention
Behavioral: Individualized counseling about both smoking cessation and weight control techniques — The FIT2 program also offers behavior coaching in diet and physical activity to restrict post-cessation weight gain, which is not covered in conventional smoking cessation services.
  Other Names: Individualized behavior coaching
  Arms: Intervention

SUMMARY:
Existing literature investigating the impact of smoking cessation on new-onset diabetes mellitus (DM) risk is conflicting.

Combing the need for smoking cessation and body weight self-management to prevent the progression of prediabetes stage into DM, with the public implementation of the second-generation cessation program, we aimed to study the effectiveness of the Fight Tobacco and Stay Fit (FIT2) program aiming at promoting smoking cessation and restricting post-cessation weight gain (PCWG) together in prediabetic smokers regarding long-term glycemic and DM-related health outcomes.

DETAILED DESCRIPTION:
Participants:

We expect to recruit study participants at National Taiwan University Hospital and its Yunlin branch, where a systematic identification system has been applied to classify the tobacco addiction status of every patient in outpatient clinics. This study invites identified current smokers to undergo screening tests between August 2013 to January 2017. All participants should give informed consent, with personal data protected. Only individuals aged 30 to 75 years are included. A history of diabetes, hypertension, Fagerström test for nicotine dependence, alcohol consumption, physical activity, depression, sleep quality, and current medications is collected through standardized personal interviews. Prediabetic participants are those who repeatedly have either of the following: 1) plasma glucose 100 to 125 mg/dL (5.6 to 6.9 mmol/L) in the fasting state; 2) plasma glucose 140 to 199 mg/dL (7.8 to 11.0 mmol/L) two hours after a 75-g oral glucose load; 3) glycosylated hemoglobin (A1C) 5.7% to 6.4%, in the absence of diabetic medications. Prediabetic participants who smoke ≥10 CPD for at least 6 months are classified as prediabetic smokers. Excluded are those with existing diagnosis of DM, thyroid diseases, acute cardiac conditions within 3 months, acute renal failure, chronic glomerulonephritis, polycystic kidney disease, mental health disorders ever diagnosed by psychiatrists, pregnancy, breast-feeding, malignancy; or current use of diabetic medications, smoking cessation medications, steroids, lithium or antipsychotics. Information about tobacco use, alcohol consumption, physical activity, depression, sleep quality, personal medical histories, and current medications is collected through standardized personal interviews and medical records. The study protocol was approved by the National Taiwan University Hospital Research Ethics Committee.

Sample size estimation We estimate to recruit at least 596 prediabetic smokers, 33% (199) of whom decide to join the intervention, to reach 90% power and a two-sided 95% CI for the detection of a 50% risk reduction, assuming 30% as the risk of incident T2D during follow-up in the usual care group.

Assignment, prospective follow-up, and analytic design The assignment of this trial is based on shared decision-making. At baseline, all eligible prediabetic smokers are asked if they would like to join the Fight Tobacco and Stay Fit (FIT2) program or just receive usual care. Beginning at enrollment, the smoking status, breath carbon monoxide levels, anthropometric indices, automated office and home blood pressures, and blood tests were recorded every six months. The intention-to-treat analysis is performed among all participants joining the FIT2 program and receiving usual care. The modified per-protocol analysis is adopted to compare participants with documented abstinence at prespecified study ends (e.g., 10 years) with the controls.

The FIT2 program and post-program abstinence:

The FIT2 program is a 16-week smoking cessation program that combines varenicline prescription with individualized counseling on not only smoking cessation but also weight control techniques. Participants in this group can receive their medications for up to 16 weeks within one year. Each participant also received counseling for individualized techniques for smoking cessation and body weight control at each visit. We do not prescribe nicotine replacement therapy (NRT) because it may induce insulin resistance and confound our study outcome. Bupropion is not available for smoking cessation in our institutions. Varenicline users are encouraged either to set their quit day 8 days after starting the medication; or to freely choose quit day at any time between Days 8 and 35 after starting treatment (i.e., following drug titration that took place within the first week). Varenicline users are also forbidden to use NRT during the study period. The varenicline prescription adheres to regulations by the Health Promotion Administration, Ministry of Health and Welfare, Taiwan (www.hpa.gov.tw) and manufacturer's directions, usually initiated at 0.5 mg once daily for the first three days and then increased to 1 mg once daily. From day 8 to up to 16 weeks, the recommended dose is 1 mg varenicline twice daily. During the therapy course, physicians are allowed to adjust varenicline dosage according to tolerability. Drug adverse events, withdrawal symptoms, and perceived barriers to quitting should be recorded and addressed. Physicians should emphasize that if there are any uncontrolled depressed moods, suicidal thoughts, or attempts, they are to cease varenicline treatment and consult a psychiatrist immediately.

Smoking status is assessed by self-reported 7-day point-prevalence abstinence, confirmed by a breath CO level. Cotinine is not used to assess abstinence because, when used with self-report to indicate whether a person has smoked, CO and cotinine levels show high agreement. We provide participants in the intervention group with individualized counseling to help minimize the relapse rate.

In addition to varenicline prescription and smoking cessation counseling covered in conventional smoking cessation services, the FIT2 program also offers individualized weekly behavior coaching in diet and physical activity to restrict PCWG. The FIT2 participants are encouraged to do at least 150 minutes of moderate-intensity (3.0-6.0 metabolic equivalents) aerobic physical activity throughout the week. The counseling sessions allow opportunities to identify obstacles to lifestyle change and to discuss approaches with a professional panel of dietitians and certified personal trainers. The FIT2 participants are encouraged to do at least 150 minutes of moderate-intensity (3.0-6.0 metabolic equivalents) aerobic physical activity throughout the week. Emphasis is placed on checking the weekly diary for body weight, food, and physical activity through protected cellphone messages between participants and the assigned panel professionals. For those who gain weight, more intensive ways of calorie restriction and physical activity (at least 300 minutes of moderate-intensity aerobic physical activity per week) are instructed.

Post-program smoking status is recorded weekly from 16 weeks to six months by self-reported 7-day point prevalence of abstinence and a breath carbon monoxide level of <6 ppm. Post-program quitters are those who quit successfully at 16 weeks after the FIT2 program and maintain their non-smoking status until the prespecified study ends (e.g., post-program abstinence at 10 years). For the modified per-protocol analysis, participants who fail to keep quit after the FIT2 program are reassigned to the control group.

Usual care and control:

Usual care is provided for prediabetic smokers who decide not to receive the FIT2 program. Usual care comprises encouragement to quit smoking and initiate a therapeutic lifestyle change at each visit. In the modified per-protocol analysis, the control group contains participants joining the FIT2 program who fail to achieve post-program abstinence and all participants receiving usual care, including those who quit smoking on their own.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 30 to 75 years
* Prediabetic smokers

Exclusion Criteria

* existing diagnosis of DM or current use of diabetic medications
* thyroid diseases
* acute cardiac conditions within 3 months
* acute renal failure, chronic glomerulonephritis, or polycystic kidney disease
* mental health disorders ever diagnosed by psychiatrists
* pregnancy or breast-feeding
* malignancy
* current use of smoking cessation medications, steroids, lithium, or antipsychotics.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 589 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2027-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hsieh Chiang, MD, MPH, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital and its Yunlin branch, Taipei, Department of Family Medicine, Taiwan

REFERENCES:
- [Background] Clair C, Rigotti NA, Porneala B, Fox CS, D'Agostino RB, Pencina MJ, Meigs JB. Association of smoking cessation and weight change with cardiovascular disease among adults with and without diabetes. JAMA. 2013 Mar 13;309(10):1014-21. doi: 10.1001/jama.2013.1644. PMID 23483176
- [Background] Bergman BC, Perreault L, Hunerdosse D, Kerege A, Playdon M, Samek AM, Eckel RH. Novel and reversible mechanisms of smoking-induced insulin resistance in humans. Diabetes. 2012 Dec;61(12):3156-66. doi: 10.2337/db12-0418. Epub 2012 Sep 10. PMID 22966072
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Cropsey KL, Eldridge GD, Weaver MF, Villalobos GC, Stitzer ML. Expired carbon monoxide levels in self-reported smokers and nonsmokers in prison. Nicotine Tob Res. 2006 Oct;8(5):653-9. doi: 10.1080/14622200600789684. PMID 17008192
- [Background] Rennard S, Hughes J, Cinciripini PM, Kralikova E, Raupach T, Arteaga C, St Aubin LB, Russ C; Flexible Quit Date Study Group. A randomized placebo-controlled trial of varenicline for smoking cessation allowing flexible quit dates. Nicotine Tob Res. 2012 Mar;14(3):343-50. doi: 10.1093/ntr/ntr220. Epub 2011 Nov 11. PMID 22080588
- [Background] Chiang CH, Yang HI, Jen CL, Lu SN, Wang LY, You SL, Su J, Iloeje UH, Chen CJ; REVEAL-HBV Study Group. Association between obesity, hypertriglyceridemia and low hepatitis B viral load. Int J Obes (Lond). 2013 Mar;37(3):410-5. doi: 10.1038/ijo.2012.63. Epub 2012 Apr 24. PMID 22531094
- [Background] Chiang CH, Lai JS, Hung SH, Lee LT, Sheu JC, Huang KC. Serum adiponectin levels are associated with hepatitis B viral load in overweight to obese hepatitis B virus carriers. Obesity (Silver Spring). 2013 Feb;21(2):291-6. doi: 10.1002/oby.20000. PMID 23404868
- [Background] Chiang CH, Lee LT, Hung SH, Lin WY, Hung HF, Yang WS, Sung PK, Huang KC. Opposite association between diabetes, dyslipidemia, and hepatocellular carcinoma mortality in the middle-aged and elderly. Hepatology. 2014 Jun;59(6):2207-15. doi: 10.1002/hep.27014. Epub 2014 Apr 3. PMID 24425422
- [Background] Chiang CH, Huang KC. Association between metabolic factors and chronic hepatitis B virus infection. World J Gastroenterol. 2014 Jun 21;20(23):7213-6. doi: 10.3748/wjg.v20.i23.7213. PMID 24966591
- [Background] Chiang CH, Huang KC. Reply: To PMID 24425422. Hepatology. 2015 May;61(5):1763-4. doi: 10.1002/hep.27427. Epub 2015 Mar 23. No abstract available. PMID 25205437
- [Background] Chang PH, Chiang CH, Ho WC, Wu PZ, Tsai JS, Guo FR. Combination therapy of varenicline with nicotine replacement therapy is better than varenicline alone: a systematic review and meta-analysis of randomized controlled trials. BMC Public Health. 2015 Jul 22;15:689. doi: 10.1186/s12889-015-2055-0. PMID 26198192
- [Background] Chiang CH, Lu CW, Han HC, Hung SH, Lee YH, Yang KC, Huang KC. The Relationship of Diabetes and Smoking Status to Hepatocellular Carcinoma Mortality. Medicine (Baltimore). 2016 Feb;95(6):e2699. doi: 10.1097/MD.0000000000002699. PMID 26871803
- [Derived] Chiang CH, Sheu YH, Guo FR, Lin WW, Chen GR, Huang KC. Incorporating Post-Cessation Weight-Control Coaching into Smoking Cessation Therapy to Reduce Type 2 Diabetes Risk. Nutrients. 2021 Sep 25;13(10):3360. doi: 10.3390/nu13103360. PMID 34684360

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention (FIT2 Program): A 16-week FIT2 program that combines smoking cessation therapy with individualized behavior coaching in diet and physical activity for PCWG restriction.
- Usual Care: Usual care is provided for prediabetic smokers who decide not to join the FIT2 program. Usual care comprises interpretation of laboratory results and encouragement to quit smoking and initiate a therapeutic lifestyle change for T2D prevention at each visit.
Period: Overall Study
Arm/Group | Intervention (FIT2 Program) | Usual Care
Started | 279 | 310
Completed | 270 | 262
Not Completed | 9 | 48

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: Usual care is provided for prediabetic smokers who decide not to join the FIT2 program. Usual care comprises interpretation of laboratory results and encouragement to quit smoking and initiate a therapeutic lifestyle change for T2 diabetes mellitus (DM) prevention at each visit.
- Total: Total of all reporting groups
Arm/Group | Intervention (FIT2 Program) | Usual Care | Total
Number analyzed (Participants) | 279 | 310 | 589
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (10.5) | 53.9 (9.4) | 53.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 51 | 98
  Male | 232 | 259 | 491
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 279 | 310 | 589
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 26.0 (3.23) | 26.4 (3.91) | 26.2 (3.61)
HbA1c [Mean (Standard Deviation); unit: percentage of HbA1c] | 6.12 (0.14) | 6.11 (0.19) | 6.11 (0.17)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With New-onset Type 2 Diabetes Mellitus (DM)
Description: The primary outcome is type 2 DM, defined as having repeatedly at least one of the following criteria: 1) plasma glucose ≥126 mg/dL (7.0 mmol/L) in the fasting state; 2) plasma glucose ≥200 mg/dL (11.1 mmol/L) randomly with hyperglycemic symptoms or two hours after a 75-g oral glucose load; 3) A1C ≥6.5%;20 or under medications for physician-diagnosed type 2 DM.
Time Frame: Up to 5 years
Population: Intention-to-treat analysis
Measure: Count of Participants; unit: Participants
Groups:
- Usual Care: Usual care comprises interpretation of laboratory results and encouragement to quit smoking and initiate a therapeutic lifestyle change for T2D prevention at each visit.
Arm/Group | Intervention (FIT2 Program) | Usual Care
Number analyzed (Participants) | 279 | 310
Participants | 83 | 134
Statistical Analysis 1: Comparison: Intervention (FIT2 Program) vs Usual Care; Test type: Superiority; p = 0.008, Regression, Cox — Statistical significance levels were determined by two-tailed tests (P < 0.05); Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.48 to 0.84]

2. Secondary Outcome: Number of Participants With Regression to Normoglycemia
Description: Participants who regress to normoglycemia should met all the following conditions for more than six months and maintained such status until the study end: 1) plasma glucose <5.6 mmol/L (100 mg/dL) in the fasting state; 2) plasma glucose <7.8 mmol/L (140 mg/dL) two hours after a 75-g oral glucose load; or 3) HbA1c<39 mmol/mol (5.7%), in the absence of antidiabetic drugs.
Time Frame: Up to 5 years
Population: Intention-to-treat analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (FIT2 Program) | Usual Care
Number analyzed (Participants) | 279 | 310
Participants | 43 | 25
Statistical Analysis 1: Comparison: Intervention (FIT2 Program) vs Usual Care; Test type: Superiority; p = 0.023, Regression, Cox — Statistical significance levels were determined by two-tailed tests (P < 0.05); Cox Proportional Hazard = 1.85, 95% CI 2-sided [1.13 to 3.04]

3. Secondary Outcome: Major Adverse Cardiac Events
Description: Cardiovascular death, non-fatal myocardial infarction, and non-fatal stroke diagnosed by specialists according to medical records
Time Frame: At 10 years (between 2022 and 2026)
Reporting Status: Not Posted, anticipated posting 2027-12

4. Secondary Outcome: Chronic Kidney Disease Progression
Description: Each participant is evaluated for the renal outcome every six months and at 10 years. Defined as progression to macroalbuminuria [urinary albumin-to-creatinine ratio (UACR), >300 mg of albumin per gram of creatinine] for ≥ 3 months, or decrease in estimated glomerular filtration rate (eGFR) to <60mL/min/1.73 m2 for ≥ 3 months, as calculated by the four-variable Modification of Diet in Renal Disease (MDRD) formula, and incident albuminuria for ≥ 3 months.
Time Frame: Every 6 months and at 10 years (between 2022 and 2026)
Reporting Status: Not Posted, anticipated posting 2027-12

5. Secondary Outcome: NAFLD Progression
Description: Each participant is evaluated for the steatohepatitic outcome using FIB-4 scores, BARD scores, liver stiffness measurement (LSM) every six months and at 10 years. A FIB-4 score <1.45 means a low risk of advanced fibrosis, whereas patients with a score >3.25 are likely to have advanced fibrosis. A BARD score of 2-4 was associated with an OR for advanced fibrosis of 17 (CI 9.2-31.9) and a negative predictive value of 96%. LSM is useful to exclude advanced NASH fibrosis with a high negative predictive value (at a cutoff <7 kPa).
  Ref: FIB-4 scores (www.mdcalc.com/fibrosis-4-fib-4-index-liver-fibrosis); BARD scores (www.mdcalc.com/bard-score-nafld-fibrosis);
Time Frame: Every 6 months and at 10 years (between 2022 and 2026)
Reporting Status: Not Posted, anticipated posting 2027-12

6. Secondary Outcome: Malignancy Incidence
Description: Incident malignancies based on medical records are accessed at 10 years, confirmed by national cancer registry system.
Time Frame: At 10 years (between 2022 and 2026)
Reporting Status: Not Posted, anticipated posting 2027-12

7. Secondary Outcome: All-Cause Mortality
Description: Deaths are ascertained at 10 years by computer linkage to the national death registry (death certificates were created by the Ministry of Health and Welfare, Taiwan) using ID numbers and these death certificates have been validated.
Time Frame: At 10 years (between 2022 and 2026)
Reporting Status: Not Posted, anticipated posting 2027-12

8. Secondary Outcome: HbA1c Change Between Baseline and 6 Months
Description: The HbA1c change (in percentage of HbA1c) was calculated from values between baseline and 6 months.
Time Frame: Baseline and 6 months
Population: Intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Intervention (FIT2 Program) | Usual Care
Number analyzed (Participants) | 279 | 310
percentage of HbA1c | 0.11 (0.15) | 0.12 (0.14)
Statistical Analysis 1: Comparison: Intervention (FIT2 Program) vs Usual Care; Test type: Other; p < 0.05, Regression, Linear; Beta Coefficient = -0.10, Standard Error of Mean 0.16

9. Other Pre Specified Outcome: 10-year Type 2 DM Risk
Description: This outcome will be collected between 2022 and 2026.
Time Frame: At 10 years
Reporting Status: Not Posted, anticipated posting 2027-12

10. Other Pre Specified Outcome: 10-year Probability of Regression to Normoglycemia
Description: This outcome will be collected between 2022 and 2026.
Time Frame: At 10 years
Reporting Status: Not Posted, anticipated posting 2027-12

11. Post Hoc Outcome: Differences Between the Automated Office and Home Blood Pressure Measurement
Description: The differences in systolic/diastolic blood pressure values (mmHg) calculated from the average automated office blood pressure (AOBP) and home blood pressure (HBP) readings are accessed every six months and at 10 years.
Time Frame: Every 6 months and at 10 years (between 2022 and 2026)
Reporting Status: Not Posted, anticipated posting 2027-12

ADVERSE EVENTS:
Time Frame: At 16 weeks and every 6 months, up to 9 years and 6 months
Arm/Group | Intervention (FIT2 Program) | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/279 | 0/310
Serious Adverse Events (participants affected / at risk) | 0/279 | 0/310
Other Adverse Events (participants affected / at risk) | 50/279 | 65/310
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (FIT2 Program) (N=279) | Usual Care (N=310)
Fatigue (General disorders) | 42 | 49
Insomnia (Psychiatric disorders) | 45 | 53

LIMITATIONS AND CAVEATS:
The selection bias could not be completely mitigated due to the allocation by shared decision-making in this study. Participants with high motivation to quit are more likely to join the FIT2 program than their counterparts. Indeed, this design conforms to pragmatic clinical practice. The use of a non-randomized control group reduces the threat to external validity, which limits the value of randomized controlled trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT01926041/Prot_SAP_000.pdf